CLINICAL TRIAL: NCT05284188
Title: The Clinical Outcomes Comparing Open and Arthroscopic Modified Broström Operation in Chronic Lateral Ankle Instability and Generalized Joint Laxity
Brief Title: The Clinical Outcomes of the Arthroscopic and Open Modified Broström Operation in CLAI and GJL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Jiang Dong, Chief physician, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2021052
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2018-01

CONDITIONS: Ankle Sprains; Instability, Joint; Joint Hypermobility
Keywords: chronic lateral ankle instability; generalized joint laxity; modified Brostrom operation; arthroscopic; open
MeSH Terms: conditions — Ankle Injuries; Joint Instability

STUDY DESIGN:
Masking Description: Randomization was achieved using the opaque sealed envelopes, and each eligible patient was allocated to open or arthroscopic MBP in a 1:1 ratio with a random block assignment of 4 or 6. The envelopes were thoroughly shuffled and sequentially numbered and then opened before surgery. Patients were allowed to withdraw from this experiment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Modified Broström operation group (Active Comparator): Patients who accept an open modified Broström operation
  Interventions: Procedure: Open or arthroscopic Modified Broström operation
- Arthroscopic Modified Broström operation group (Active Comparator): Patients who accept an arthroscopic modified Broström operation
  Interventions: Procedure: Open or arthroscopic Modified Broström operation

INTERVENTIONS:
Procedure: Open or arthroscopic Modified Broström operation — Patients with CLAI and GJL were randomly allocated to accept the open or arthroscopic Modified Broström operation.

SUMMARY:
Investigators designed this randomized controlled trial to compare the clinical outcomes of open and arthroscopic modified Broström operation for the treatment of CLAI and GJL.

DETAILED DESCRIPTION:
The open modified Broström operation is the first line to treat chronic lateral ligament instability (CLAI). Arthroscopic techniques gain popularity for less invasivity, quick recovery to normal and sports activities, and the possibility to treat other intraarticular disorders. Studies have shown significantly poor clinical and radiological outcomes and a higher rate of failure in patients with generalized joint laxity (GJL) than patients without after open modified Broström operation. However, there is no study to compare the open and arthroscopic modified Brostrom operation for patients with GJL and CLAI. So, investigators designed this randomized controlled trial. The primary outcomes are Karlsson, American Orthopaedic Foot & Ankle Society, and visual analogue scales. The secondary outcomes are anterior displacement and talar tilt angle in stress radiography, the rate of re-injury.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of lateral ankle pain and instability Beighton score ≥4 Age with 18 to 60 years

Exclusion Criteria:

- Patients with an acute or subacute ankle injury (within 3 months) Injury of the deltoid ligament Alignment of lower extremity greater than 5 degrees Fractures of the lower extremity Stage III or IV osteoarthritis Patients who refused to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Karlsson score | postoperative Karlsson score at 1 year
  This score is a primary scale for lateral ankle instability
Karlsson score | postoperative Karlsson score at 2 years
  This score is a primary scale for lateral ankle instability

SECONDARY OUTCOMES:
Anterior displacement and talar tilt angle in stress radiography | postoperative radiographic measures at 2 years
  The outcomes are common indicators for evaluation the lateral stability of ankle

CONTACTS AND LOCATIONS:
Overall Officials: Dong Jiang, MD, Principal Investigator — Peking University Third Hosptial
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
The demographics data, Beighton score, primary and secondary outcomes would be available to other researchers

REFERENCES:
- [Background] de Vries JS, Krips R, Sierevelt IN, Blankevoort L, van Dijk CN. Interventions for treating chronic ankle instability. Cochrane Database Syst Rev. 2011 Aug 10;(8):CD004124. doi: 10.1002/14651858.CD004124.pub3. PMID 21833947
- [Background] Sacks HA, Prabhakar P, Wessel LE, Hettler J, Strickland SM, Potter HG, Fufa DT. Generalized Joint Laxity in Orthopaedic Patients: Clinical Manifestations, Radiographic Correlates, and Management. J Bone Joint Surg Am. 2019 Mar 20;101(6):558-566. doi: 10.2106/JBJS.18.00458. No abstract available. PMID 30893238
- [Background] Xu HX, Lee KB. Modified Brostrom Procedure for Chronic Lateral Ankle Instability in Patients With Generalized Joint Laxity. Am J Sports Med. 2016 Dec;44(12):3152-3157. doi: 10.1177/0363546516657816. Epub 2016 Aug 5. PMID 27496909
- [Background] Park KH, Lee JW, Suh JW, Shin MH, Choi WJ. Generalized Ligamentous Laxity Is an Independent Predictor of Poor Outcomes After the Modified Brostrom Procedure for Chronic Lateral Ankle Instability. Am J Sports Med. 2016 Nov;44(11):2975-2983. doi: 10.1177/0363546516656183. Epub 2016 Aug 1. PMID 27480980
- [Background] Li H, Hua Y, Li H, Ma K, Li S, Chen S. Activity Level and Function 2 Years After Anterior Talofibular Ligament Repair: A Comparison Between Arthroscopic Repair and Open Repair Procedures. Am J Sports Med. 2017 Jul;45(9):2044-2051. doi: 10.1177/0363546517698675. Epub 2017 Apr 10. PMID 28394631
- [Derived] Wang AH, Su T, Jiang YF, Zhu YC, Jiao C, Hu YL, Guo QW, Jiang D. Arthroscopic modified Brostrom procedure achieved similar favorable short term outcomes to open procedure for chronic lateral ankle instability cases with generalized joint laxity. Knee Surg Sports Traumatol Arthrosc. 2023 Sep;31(9):4043-4051. doi: 10.1007/s00167-023-07431-x. Epub 2023 May 10. PMID 37162539